CLINICAL TRIAL: NCT02380976
Title: Phase 1 Clinical Trial of DW340 and DW330SR + DW1030 Co-administration in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW340-1002
Record Dates: First submitted 2015-02-24; First posted 2015-03-05 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Healthy

ARMS (2):
- Test 1 (Experimental): First phase: DW330SR+DW1030 7 days after Second phase: DW340
  Interventions: Drug: combination drug: DW330SR, DW1030; Drug: DW340
- Test 2 (Experimental): First phase: DW340 7 days after Second phase: DW330SR+DW1030
  Interventions: Drug: combination drug: DW330SR, DW1030; Drug: DW340

INTERVENTIONS:
Drug: combination drug: DW330SR, DW1030
Drug: DW340

SUMMARY:
A randomized, open-label, single-dose, crossover Phase I Study to investigate the relative bioavailability of DW340 and DW330SR + DW1030 co-administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age at screening visit only 20 healthy men over the age of 40 years or less
* Screening visit, BMI measurement is more than 19 kg/m2 who are below 27 kg/m2
* Screening vist, 90 mmHg ≤ SBP ≤ 140 mmHg, 50 mmHg ≤ DBP ≤ 90 mmHg
* Fully understand the purpose of trial, test drug and follow the instructions of the trial, Those who voluntarily written consent that ability and decision to participate during the entire period of the test

Exclusion Criteria:

* Those with a clinically significant history or character; Liver, kidney, digestive, respiratory, musculoskeletal, endocrine, neuropsychiatric, blood • tumor type, cardiovascular disease
* Those with Gastrointestinal diseases that may affect the absorption of the IND or history of surgery
* Those who have a clinically significant history of hypersensitivity to drug and food
* Those with genetic problems, such as galactose intolerance, lactase deficiency or glucose-galactose malabsorption
* Within 60 days those taking the other clinical trial drug
* Within 30 days those who take the drug metabolizing enzyme induction and inhibition drugs or prescription drugs
* Within 30 days those who take food abnormally, that may affect ADME of drug
* Within 60 days those who donate whole blood, within 30 days those who donate blood partially, receive transfusion
* Within 14 days those who take OTC drug
* Those who showing positive for drug abuse concerns in urine drug testing
* Those who drink excessive alcohol or have history of alcoholism
* Heavy smoker
* and so on

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cmax of DW330SR | 9 days
Cmax of DW340 | 9 days
Cmax of DW1030 | 9 days
AUClast of DW330SR | 9 days
AUClast of DW340 | 9 days
AUClast of DW1030 | 9 days